CLINICAL TRIAL: NCT06848166
Title: Study of the Effectiveness and Safety of Embolization of the Middle Meningeal Artery Using Non-adhesive Materials SQUID 12 and SQUID 18 in the Treatment of Patients With Chronic Resistant Migraine
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vedanta University Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MigraSquid1812
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Chronic Migraine Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with chronic resistant migraine (Experimental)
  Interventions: Device: liquid embolic agent SQUID 12, liquid embolic agent SQUID 18

INTERVENTIONS:
Device: liquid embolic agent SQUID 12, liquid embolic agent SQUID 18 — Total endovascular embolization of the frontal and parietal branches (less often the occipital branch) of the middle meningeal artery (MMA) with its complete devascularization. In the case of unilateral pain localization, ipsilateral MMA embolization will be performed; in the case of bilateral pain localization, total embolization of both MMA branches will be performed.

SUMMARY:
To evaluate the effectiveness and safety of middle meningeal artery (MMA) embolization using non-adhesive materials SQUID 12 and SQUID 18 as a treatment method for patients with chronic resistant migraine.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has read, understood, signed, and dated the Patient Information Sheet with the informed consent form.
2. The patient is aged between 35 and 59 years inclusive at the time of signing the Patient Information Sheet with the informed consent form.
3. The diagnosis of "chronic migraine" according to the clinical guidelines on migraine by the Ministry of Health of the Russian Federation (2021) / ICD-10 (2018), established at least 12 months before screening.
4. Resistant nature of the migraine, determined by the doctor using the criteria of the European Headache Federation (EHF, 2020), established at least 6 months before screening.
5. At least 14 days of headache during the screening period (28 days), of which 8 days of headache meet the definition of migraine (assessed based on the results of filling out the Headache Diary for 28 days during the screening period).
6. Migraine, resistant to both pharmacological and non-pharmacological prevention and treatment methods, in the patient's history.
7. Maximum level of headache during migraine days above 5 points (inclusive) on a 10-point numerical rating scale during the screening period.
8. No positive effect on migraine symptoms (frequency and intensity of headache attacks) from previous botulinum toxin therapy (administration of OnabotulinumtoxinA, Relatox® (botulinum toxin type A - hemagglutinin complex 155 - 195 IU, administered every 12 weeks according to the PREEMPT protocol).
9. Consent to use adequate contraceptive methods* and not serve as an egg/sperm donor from the time of signing the Patient Information Sheet with the informed consent form for participation in the study until the end of the study (for women with reproductive potential and men).

Exclusion Criteria:

1. The patient has contraindications to undergoing embolization of the middle meningeal artery based on the medical history, results of examinations, and laboratory tests conducted during screening.
2. Allergic reactions to contrast agents used during procedures before/during the embolization procedure and associated procedures.
3. The patient has a history of cerebral vascular malformations, arteriovenous malformations, brain aneurysms, brain tumors, hydrocephalus, arachnoiditis, cerebrospinal fluid circulation disorders, craniovertebral junction anomalies, platybasia, skull base deformities, severe traumatic brain injuries, stenosis, and occlusion of pre-cerebral arteries.
4. The patient has a history of skull base fractures and consequences of skull base fractures, history of neurosurgical operations.
5. A history of mental illness (including depression, confirmed by a psychiatrist during screening through the HADS questionnaire and Hamilton scale assessment), which, in the opinion of the psychiatrist, may affect the patient's ability to assess their condition, interfere with participation in the study, or impact the patient's safety during the study.
6. A history of hyperthyroidism or diabetes. The presence of other endocrine disorders in the patient's history that, in the doctor's opinion, could interfere with participation in the study or affect the evaluation of efficacy and/or safety.
7. History or data of drug addiction, alcoholism, or abuse of medications.
8. Medication-induced headache at the time of screening and within 3 months (12 weeks) prior to screening.
9. Other types of chronic headache in the patient's history within less than 12 months before screening, such as trigeminal autonomic cephalalgias (including cluster headaches, prolonged hemicrania), new daily persistent headaches, painful cranial neuropathies, retinal migraine, aura without headache, hemiplegic migraine, brainstem aura migraine, idiopathic intracranial hypertension without optic nerve edema, spontaneous intracranial hypertension, secondary headaches.
10. The patient is unable to distinguish a migraine headache from other types of headache.
11. The patient has migraine complications, such as status migrainosus, persistent aura without infarction, migraine infarction, migraine aura (as a trigger for epileptic seizures).
12. Body mass index (BMI) below 18.5 or above 39.9 kg/m².
13. The onset of migraine was diagnosed at an age older than 50 years.
14. The presence of metabolic syndrome or cachexia.
15. Severe cardiovascular diseases currently or in the past, including: chronic heart failure class III or IV (according to the New York Heart Association classification), clinically significant ventricular arrhythmias (ventricular tachycardia, ventricular fibrillation), significant heart valve diseases, uncontrolled hypertension with systolic blood pressure > 180 mm Hg and diastolic blood pressure > 110 mm Hg, pulmonary embolism, or deep vein thrombosis.
16. Varicose veins of the lower limbs, history of lower limb vein thrombosis.
17. Ischemic heart disease, atherosclerosis of coronary vessels.
18. Stenotic atherosclerosis of brachiocephalic arteries in the patient's history.
19. Acute cerebrovascular accident or its consequences in the patient's history.
20. The patient is pregnant or plans to become pregnant within the next 3 months.
21. Atrial fibrillation, patent foramen ovale, anomalies of the interatrial septum, history of heart and coronary vessel surgeries.
22. Signs of blood clotting disorders in the patient's history and screening, history of antiphospholipid syndrome.
23. Use of anticoagulant drugs less than 5 days before the procedure.
24. Uncontrolled bronchial asthma, severe chronic obstructive pulmonary disease in the patient's history.
25. Renal insufficiency at screening based on the calculation of glomerular filtration rate (GFR) ≤ 60 mL/min, based on serum creatinine levels at screening, or a history of renal insufficiency.
26. History of liver insufficiency, elevated ALT and AST levels at screening.
27. History of generalized pain syndrome, fibromyalgia.
28. For women: use of combined oral contraceptives with a history of thrombosis of any localization.
29. History of epilepsy, epileptic syndrome, seizure disorders, neurological conditions other than the primary condition (migraine).
30. Presence of antibodies to HIV, hepatitis C virus, hepatitis B surface antigen (HbsAg), antibodies to T. Pallidum, or a history of HIV infection, hepatitis B, hepatitis C, or syphilis, either in the medical history or based on the results of serological blood tests at screening.
31. Malignant neoplasms within 5 years before screening, or current or suspected oncological disease.
32. Other serious, unstable, decompensated, or clinically significant medical or psychological conditions that, in the opinion of the doctor, may interfere with the patient's participation in the study or affect the evaluation of efficacy and/or safety.
33. Participation in other interventional clinical trials, including the study completion visit, within 30 days prior to the screening, or planning to participate in such studies during the current study. Participation in non-interventional registry or epidemiological studies is allowed.
34. The patient is unable to read or write, unwilling or unable to comply with the study protocol procedures; any other conditions that, in the opinion of the doctor, may prevent participation in the study, adherence to procedures, or contradict the patient's interests, as well as affect the study results.
35. Employees of the medical institution conducting the study or the sponsor company, their family members, or subjects in dependent relationships.

Ages: 35 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
number of migraine days | From previous 4 weeks before enrollment to the 3 months (12 weeks) post-surgery
  Change from baseline (during the screening period) in the number of migraine days over the previous 4 weeks, assessed at 3 months (12 weeks) post-surgery

SECONDARY OUTCOMES:
The number of migraine days after surgery | From surgery up to 1 month (4 weeks), 2 months (8 weeks), 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) post-surgery
  The number of migraine days over the previous 4 weeks at 1 month (4 weeks), 2 months (8 weeks), 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) post-surgery
The average number of migraine days | From treatment every 12-week period, assessed at visits 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) post-surgery
  The average number of migraine days over a 4-week period, calculated for the preceding 12-week period, assessed at visits 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) post-surgery
Change from baseline (during the screening period) in the number of migraine days over the previous 4 weeks, assessed at 1 month (4 weeks), 2 months (8 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) post-surgery. | From screening up to 12 months
  Change from baseline (during the screening period) in the number of migraine days over the previous 4 weeks, assessed at 1 month (4 weeks), 2 months (8 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) post-surgery.
The number of headache days over the previous 4 weeks at 1 month (4 weeks), 2 months (8 weeks), 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) post-surgery | From surgery up 12 months (48 weeks) post-surgery
  The number of headache days over the previous 4 weeks at 1 month (4 weeks), 2 months (8 weeks), 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) post-surgery
The average number of headache days over a 4-week period, calculated for the preceding 12-week period, assessed at visits 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) post-surgery. | From surgery up 12 months (48 weeks) post-surgery
  The average number of headache days over a 4-week period, calculated for the preceding 12-week period, assessed at visits 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) post-surgery.
Change compared to the baseline level (during the screening period) of the number of days with headaches in the previous 4 weeks, assessed at 1 month (4 weeks), 2 months (8 weeks), 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 | From screening up to 12 months
  Change compared to the baseline level (during the screening period) of the number of days with headaches in the previous 4 weeks, assessed at 1 month (4 weeks), 2 months (8 weeks), 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) after the surgery.
The proportion of patients whose number of migraine days in the previous 4 weeks decreases by 50% or more from the baseline level | From surgery up 12 months (48 weeks) post-surgery
  The proportion of patients whose number of migraine days in the previous 4 weeks decreases by 50% or more from the baseline level (during the screening period) at 1 month (4 weeks), 2 months (8 weeks), 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) after the surgery.
The proportion of patients whose average number of migraine days over the previous 12 weeks decreases by 50% or more | From screening up to 12 months
  The proportion of patients whose average number of migraine days over the previous 12 weeks decreases by 50% or more at the visit at 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) after the surgery, compared to the baseline level (during the screening period).
The proportion of patients whose number of headache days in the previous 4 weeks decreases by 50% or more from the baseline level | From screening up to 12 months
  The proportion of patients whose number of headache days in the previous 4 weeks decreases by 50% or more from the baseline level (during the screening period) at 1 month (4 weeks), 2 months (8 weeks), 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) after the surgery.
The number of days with headache intensity rated as "moderate" or "severe" in the previous 4 weeks | From surgery up 12 months (48 weeks) post-surgery
  The number of days with headache intensity rated as "moderate" or "severe" in the previous 4 weeks at 1 month (4 weeks), 2 months (8 weeks), 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) after the surgery (according to the Clinical Trial Guidelines for Chronic Migraine Prevention, 2018).
The average number of days in the previous 12-week period with headache intensity rated as "moderate" or "severe," | From surgery up 12 months (48 weeks) post-surgery
  The average number of days in the previous 12-week period with headache intensity rated as "moderate" or "severe," calculated and assessed at visits at 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) after the surgery.
Change compared to the baseline level in the number of days with headache intensity rated as "moderate" or "severe" in the previous 4 weeks | From surgery up 12 months (48 weeks) post-surgery
  Change compared to the baseline level in the number of days with headache intensity rated as "moderate" or "severe" in the previous 4 weeks, calculated at 1 month (4 weeks), 2 months (8 weeks), 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) after the surgery.
The maximum intensity of migraine headache in the previous 4 weeks, as determined by the patient using a 10-point numerical rating scale | From surgery up 6 months (24 weeks) post-surgery
  The maximum intensity of migraine headache in the previous 4 weeks, as determined by the patient using a 10-point numerical rating scale, assessed at 1 month (4 weeks), 2 months (8 weeks), 3 months (12 weeks), and 6 months (24 weeks) after the surgery.
The number of days with symptoms associated with migraine (nausea, vomiting, photophobia, phonophobia) in the previous 4 weeks | From surgery up 6 months (24 weeks) post-surgery
  The number of days with symptoms associated with migraine (nausea, vomiting, photophobia, phonophobia) in the previous 4 weeks, assessed at 1 month (4 weeks), 2 months (8 weeks), 3 months (12 weeks), and 6 months (24 weeks) after the surgery.
The total score on the HIT-6 scale | From surgery up 12 months (48 weeks) post-surgery
  The total score on the HIT-6 scale at 1 month (4 weeks), 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) after the surgery.
The total score on the MIDAS scale | From surgery up 12 months (48 weeks) post-surgery
  The total score on the MIDAS scale at 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) after the surgery.
Change in the total score on the HIT-6 scale | From surgery up 12 months (48 weeks) post-surgery
  Change in the total score on the HIT-6 scale at 1 month (4 weeks), 2 months (8 weeks), 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), and 12 months (48 weeks) after the surgery compared to the baseline level.

CONTACTS AND LOCATIONS:
Overall Officials: Andrey S Petrov, MD, PhD, Principal Investigator — Vedanta Clinic
Locations (1):
- Vedanta University Clinic, Bishkek, Gorod Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided
Decision on IPD sharing is in progress